CLINICAL TRIAL: NCT06695611
Title: Evaluating the Feasibility of a Randomized Cluster Trial for Blood Pressure Targets in In-centre Hemodialysis Units (BP in HD Pilot Trial)
Brief Title: Feasibility of a Randomized Cluster Trial for Blood Pressure Targets in In-centre Hemodialysis Units
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Navdeep Tangri, Principal Investigator/Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS26418 (B2024:040)
Record Dates: First submitted 2024-10-28; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Disease 5D
Keywords: Chronic Kidney Diseases; Blood Pressure; End Stage Renal Disease; Hemodialysis; Dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: This pilot study is a 4-centre pragmatic, two-arm, parallel-group, open-label cluster-randomized trial evaluating the feasibility of implementing a higher versus lower blood pressure target protocol
Who Masked: Outcomes Assessor
Masking Description: As this is an open-label cluster randomization, the unit staff and patients will be aware of their unit's target blood pressure. The statistician performing the data analysis will be blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Higher pre-dialysis blood pressure target (150-170 mm Hg systolic) (as a unit-level policy) (Active Comparator): The approach to reach blood pressure target is up to the treating physician. Depending on baseline pre-dialysis systolic blood pressure, blood pressure may need to be raised or lowered to reach the target.
  Interventions: Other: Increase systolic blood pressure; Other: Decrease systolic blood pressure
- Lower pre-dialysis blood pressure target (110-140 mm Hg systolic) (as a unit-level policy) (Experimental): The approach to reach blood pressure target is up to the treating physician. Depending on baseline pre-dialysis systolic blood pressure, blood pressure may need to be raised or lowered to reach the target.
  Interventions: Other: Increase systolic blood pressure; Other: Decrease systolic blood pressure

INTERVENTIONS:
Other: Increase systolic blood pressure — To increase systolic blood pressure, treating physicians can consider the following options:
  1. Withdraw blood pressure medications, reducing dose of medications that are not indicated for other reasons, or down titrate medication.
  2. Increase estimated dry weight (EDW) by 0.5 kg increments if the participant is hypovolemic or euvolemic
Other: Decrease systolic blood pressure — To decrease SBP, treating physicians can consider the following options:
  1. Adjust blood pressure medications. This could be accomplished by increasing the dose of current medications, and/or adding an additional medication class. Choice of medication will be dependent on current medications, contraindications, age, comorbidities, and cardiovascular indications. Adherence to blood pressure medications should be reviewed.
  2. Reduce EDW by 0.1 - 0.5 kg
  3. Reduce sodium levels. This could be accomplished through a reduction in dietary sodium intake to <2 gm/day and fluid intake to <1.5 L per day. Adherence to dietary sodium restrictions should be reviewed with the participant
  4. Extend dialysis time or adding an additional dialysis session if needed to achieve target dry weight

SUMMARY:
High blood pressure in people receiving hemodialysis is known to contribute to heart disease and heart-related death from strokes, heart failure, left ventricular hypertrophy (which is a thickening of the heart wall that makes it difficult for the heart to pump blood) and arrythmias (an irregular or abnormal heartbeat). In comparison, low blood pressure can lead to cramps, myocardial stunning, and cerebrovascular ischemia. However, despite, blood pressure management being an important component of hemodialysis care, the "best" blood pressure target for people on hemodialysis is unknown.

Finding the "right" blood pressure to target can have a major impact on patient lives. We are proposing a large, pragmatic, cluster randomized trial targeting a lower versus higher blood pressure target in in-centre hemodialysis units in Canada. Our initial steps towards this bigger trial are to run a smaller trial including 4 units, to evaluate whether it is feasible to conduct a larger trial. Our ultimate goal is to deliver the definitive randomized trial for blood pressure targets in the hemodialysis population.

DETAILED DESCRIPTION:
Despite, blood pressure management being a cornerstone of multidisciplinary rounds, the optimal blood pressure target for people on hemodialysis is unknown. We plan to conduct a pilot study to determine if implementation of a pre-dialysis blood pressure protocol (as a unit-level policy) of a higher (150-170 mm Hg systolic) versus lower target (110-140 mm Hg systolic) in patients receiving chronic, in-centre hemodialysis is feasible?

This pilot study is a 4-centre pragmatic, two-arm, parallel-group, open-label cluster-randomized trial evaluating the feasibility of implementing a higher versus lower blood pressure target protocol. The intervention period will last 3 months, with check-ins at weeks 4 and 8 to see if clusters are able to meet their target blood pressures. If blood pressures are not at target at the week 4 check-in, a review between the study team and cluster will be conducted to determine how the target can be achieved.

Clusters will be randomized to a target pre-dialysis SBP of 110-140 mm Hg (the treatment arm) or 150-170 mm Hg (the standard arm). A 2-week average of standardized pre-dialysis systolic blood pressure readings measured in unknit will be used to define blood pressure targets and goals. Two weeks after a change to treatment has been made, SBP should be reassessed. If it is still above or below target range, another adjustment to course of treatment should be made. This interval allows for the effects of the change in treatment to be seen before any additional changes in treatment are made. The decision on how to adjust a participant's treatment in order to meet target blood pressure is up to the treating physician. This allows for more flexibility in treatment options and greater individuality in care. The treating physician can make treatment decisions based on individual needs, so as to better account for the participant's counter indication, comorbidities, and tolerances. Significant changes (both increases and decreases) in dry weight are not recommended. Changes in anti-hypertensive medication titration is the preferred option to adjust blood pressure before adjusting dry weight, sodium, and dialysis time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Undergoing in-centre hemodialysis at least twice weekly
* > 90 days since initiation of dialysis

Exclusion Criteria:

* Participation in another intervention study that may affect blood pressure other than other cluster RCTs of dialysate composition
* Inability to measure blood pressures in an upper arm
* Pregnancy, anticipated pregnancy, or breastfeeding
* Unmeasurable SBP (e.g., have left ventricular assist device)
* Life expectancy < 4 months
* Planned transition to home dialysis within 3 months
* Planned move to a different dialysis unit within 3 months
* Anticipated living donor kidney transplant within 3 months
* Other reasons as determined by treating clinician, reasons will be recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference in blood pressure between arms | Week 11 to13
  Difference in 2-week average (week 11 to13) pre-dialysis SBP between treatment arms

SECONDARY OUTCOMES:
Feasibility Outcomes - Proportions | Week 13
  1. The proportion of patients who reach target
  2. The proportion of patients declined changing their prescribed SBP target
  3. The proportion of patients for whom a care provider did not agree to changing the prescribed SBP target
Feasibility Outcomes - Change since baseline | Baseline and week 13
  Change in dry weight
Incidence of Adverse Events | Week 13
  1. Number of recorded cramps
  2. Requirement for fluid bolus
  3. SBP <90 or > 200 mm Hg requiring intervention
  4. Hospitalizations or ER visits related to fluid overload
  5. Dizziness, falls, or syncope
  6. Vascular access thrombosis
  7. Major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Navdeep Tangri, MD, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data comes from chart reviews and will not be shared.